CLINICAL TRIAL: NCT01042340
Title: Energy Dense Oleic Acid Rich Formula to Newly Admitted Geriatric Patients - Feasibility and Effects on Energy Intake
Brief Title: Energy Dense Oleic Acid Formula to Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Gerd Faxén Irving, Karolinska University Hosptial Huddinge and Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Karolinska University Hospital
Record Dates: First submitted 2009-12-30; First posted 2010-01-05 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2009-12

CONDITIONS: Nutritional Intervention
Keywords: nutrition; geriatric; supplement; energy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention with energy dense formula (Experimental): Patients were randomised to intervention with the energy dense formula Calogen.
  Interventions: Other: Calogen® - an energy dense oleic acid based formula
- Control group (No Intervention): The patients that were randomised to control group were assigned to ordinary treatment.

INTERVENTIONS:
Other: Calogen® - an energy dense oleic acid based formula — A daily dose of 3 x 30 ml of Calogen®, strawberry flavour, distributed at the same time as the pharmaceutical prescriptions, i.e. at 7.00, 14.00 and 20.00.
  Other Names: SHS International LTD, UK; Nutricia Nordica AB, Sweden
  Arms: Intervention with energy dense formula

SUMMARY:
Background and aims:

Old patients seldom reach energy requirements. The effects of an oleic-acid rich formula on energy intake and appetite were studied.

Methods: Recently admitted geriatric patients (n=71), likely to stay more than 1 week were randomised to receive a fat emulsion (Calogen, intervention group (IG)) or to standard care (control group (CG)). Thirty ml of the emulsion were given 3 times daily, i.e. 420 kcal, and was distributed at the regular medication rounds. Food intake and self-rated appetite were registered 2-3 days after admission and on day 8 or the day prior to discharge. Nutritional risk screening (NRS) 2002 and serum lipids and fatty acid profiles were analysed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: likely to stay at the ward more than one week, >65 years old and able to give informed consent.

Exclusion Criteria:

* Exclusion criteria were: pancreatitis, fat malabsorption, overweight (BMI >30) and non-consent for participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To detect a significant difference in energy intake of 48kJ/200 kcal between the groups at 5% significance level and with 80% power. | 5 days to 3 weeks intervention

SECONDARY OUTCOMES:
Effects on serum lipids and appetite | 5 days to 3 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Faxén Irving, PhD, Principal Investigator — Dep of Clinical Nutrition and dietetics Karolinska University Hospital and section of Clinical Nutrition/NVS/Karolinska Institute
Locations (1):
- Dep of Geriatrics, Karolinska University Hospital, Huddinge, Stockholm, Sweden

REFERENCES:
- [Background] Milne AC, Potter J, Avenell A. Protein and energy supplementation in elderly people at risk from malnutrition. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003288. doi: 10.1002/14651858.CD003288.pub2. PMID 15846655
- [Derived] Faxen-Irving G, Cederholm T. Energy dense oleic acid rich formula to newly admitted geriatric patients--feasibility and effects on energy intake. Clin Nutr. 2011 Apr;30(2):202-8. doi: 10.1016/j.clnu.2010.08.007. Epub 2010 Sep 19. PMID 20855136